CLINICAL TRIAL: NCT00368264
Title: A Double Blind, Randomized, Placebo Controlled, Multi-Center Trial of Anti-TNF-alpha Chimeric Monoclonal Antibody (Infliximab) and Azathioprine in Patients Suffering From Systemic Lupus Erythematosus (SLE) With WHO Class V Glomerulonephritis
Brief Title: TNF Blockade With Remicade in Active Lupus Nephritis WHO Class V (TRIAL )
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Failure to recruit patients with membranous lupus nephritis not previously treated with azathioprine .
Sponsor: Medical University of Vienna (Other)
Collaborators: Hospital Hietzing (Other); Medical University of Graz (Other); Charite University, Berlin, Germany (Other); University of Erlangen-Nürnberg (Other); Heinrich-Heine University, Duesseldorf (Other); University Medical Center Groningen (Other); Leiden University Medical Center (Other); Radboud University Medical Center (Other)
Responsible Party: Prof. Josef S. Smolen, Head, Department of Medicine III, Department of Medicine III, Medical University of Vienna, Austria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRIAL V; Eudract-Nr. 2005-004067-30; Protocol EU-116; EK Nr:110/2006
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2009-10-05 (Estimated); Status verified 2009-10

CONDITIONS: Lupus Erythematosus, Systemic; Lupus Nephritis
Keywords: lupus; nephritis; membraneous; proteinuria; TNF; infliximab; azathioprine; autoantibodies
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis; Nephritis; Proteinuria | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Experimental): azathioprine plus 4 infusions of infliximab (5 mg/kg)
  Interventions: Drug: infliximab
- 2 (Placebo Comparator): azathioprine plus 4 placebo infusions
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: infliximab — azathioprine (2 mg/lkg) plus four infusions of infliximab (5mg/kg)
  Arms: 1
Drug: placebo — azathioprine (2 mg/kg) plus four placebo infusions
  Arms: 2

SUMMARY:
Background:

Standard therapy is ill-defined for patients with systemic lupus erythematosus (SLE) suffering from the membraneous form of Lupus nephritis (WHO class V). Therapeutic options used at present include azathioprine.

In a small, open label safety study, patients with lupus nephritis, including patients with membraneous lupus nephritis, have experienced a long-lasting therapeutic response, with sustained reduction in proteinuria, following a 10 weeks course of 4 infusions of infliximab in combination with azathioprine. This short course appeared safe with regard to SLE activity, despite increases in autoantibody levels.

Study hypothesis:

1. The combination of four infusions of infliximab (5 mg/kg of body weight)administered at weeks 0, 2,6, and 10, with azathioprine will be faster than azathioprine alone in reducing proteinuria to less than 1.5 g/day in patients with active lupus nephritis WHO class V (proteinuria > 3g/day).
2. This combination therapy will show a tolerable safety profile with regard to SLE activity and infections.

ELIGIBILITY:
Inclusion Criteria:

* SLE (ACR criteria fulfilled) with biopsy-proven membranous glomerulonephritis (WHO class V).
* Proteinuria > 3 g/day despite adequate therapy with ACE inhibitors and steroids (at least 2 months treatment with steroids with a dose at any time of at least 50 mg prednisolone (or equivalent), and ACE inhibitors and/or AT II antagonists at their maximum daily dose or, if this cannot be reached, the maximum daily dose tolerated).
* Capacity to understand and sign an informed consent form.
* Men and women of childbearing potential must use adequate birth control measures for the duration of the study and should continue such precautions for 6 months after receiving the last infusion.
* No history of latent or active TB prior to screening.
* No signs or symptoms suggestive of active TB upon medical history and/or physical examination.
* No recent close contact with a person with active TB or, if there has been such contact, will be referred to a physician specializing in TB to undergo additional evaluation and, if warranted, receive appropriate treatment for latent TB prior to or simultaneously with the first administration of study agent.
* Within 1 month prior to the first administration of study agent, either have a negative tuberculin skin test, or have a newly identified positive tuberculin skin test during screening in which active TB has been ruled out and for which appropriate treatment for latent TB has been initiated either prior to or simultaneously with the first administration of study agent.
* Have a chest radiograph (both posterior-anterior and lateral views) with no evidence of current active TB or old inactive TB.
* Screening laboratory test results meet the following criteria:

  * WBC (white blood cell count): > 3.0 109/L
  * Hemoglobin: > 6 mmol/L (9,6 g/dL)
  * Platelets: 100-350 109/L
  * Serum Creatinine: 1.5 times the upper limit of normal range
  * ALAT / ASAT within twice the upper normal range.

Exclusion Criteria:

* Active WHO class IV SLE nephritis.
* Treatment with Azathioprine within the previous 12 months.
* Treatment with cyclophosphamide within the previous 12 months.
* Treatment with cyclosporine within the previous 6 weeks.
* Active cerebral SLE
* Presence of anti-phospholipid-antibodies unless under adequate anticoagulation
* Women who are pregnant, nursing, or planning pregnancy within 6 months after the last infusion.
* Have had any previous treatment with monoclonal antibodies or antibody fragments.
* History of receiving human/murine recombinant products or a known allergy to murine products. A known allergy to murine product is definitely an exclusion criterion
* Documentation of seropositive for human immunodeficiency virus (HIV).
* A positive test for hepatitis B surface antigen or hepatitis C.
* Alcohol or substance abuse
* Known history of serious infections in the previous 3 months.
* Opportunistic infection within 6 months prior to screening.
* History of latent or active granulomatous infection.
* Bacille Calmette-Guerin (BCG) vaccination within 12 months of screening.
* Chest radiograph within 3 months prior to randomization suggestive of malignancy or current active infection.
* Nontuberculous mycobacterial infection or opportunistic infection within 6 months prior to screening.
* History of lymphoproliferative disease.
* Any known malignancy or history of malignancy within the previous 5 years, with the exception of basal cell or squamous cell carcinoma of the skin that has been fully excised with no evidence of recurrence.
* Current signs or symptoms of severe, progressive or uncontrolled renal (other than disease under investigation), hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease.
* Use of any investigational drug within 30 days prior to screening or within 5 half-lives of the investigational agent, whichever is longer.
* Previous treatment with drugs targeted at reducing TNF.
* Presence of a transplanted solid organ (with the exception of a corneal transplant > 3 months prior to screening).
* Concomitant diagnosis or history of congestive heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Comparison of time needed to reduce proteinuria to 1.5 g/day or less between the infliximab plus azathioprine and the azathioprine only group.

SECONDARY OUTCOMES:
Percentage of patients reaching reduction in proteinuria to ≤ 1.5 g/day, at week 12 and week 52.
Percent reduction in proteinuria at 6 weeks, 12 weeks, 20 weeks, 36 weeks, and 52 weeks after the first infusion.
Absolute reduction in proteinuria at 6 weeks, 12 weeks, 20 weeks, 36 weeks, and 52 weeks after the first infusion.
Percent reduction in protein/ creatinine ratio.
Percent reduction in SLE disease activity (measured by SIS and SLEDAI).
Absolute reduction in SLE disease activity (measured by SIS and SLEDAI).
Changes in Quality of life as determined by the SF36 questionnaire.
Changes in Fatigue as determined by the FSS (Fatigue Severity Scale).

CONTACTS AND LOCATIONS:
Overall Officials: Josef S Smolen, MD, Study Chair — Head, Department of Rheumatology, Internal Medicine III, Medical University of Vienna, Austria; Martin Aringer, MD, Principal Investigator — Department of Rheumatology, Internal Medicine III, Medical University of Vienna, Austria; Falk Hiepe, MD, Principal Investigator — Rheumatology, Charite, Berlin, Germany; Marc Bijl, MD, Principal Investigator — Clinical Immunology, Groningen University Hospital, Netherlands
Locations (9):
- Austria (3):
  - Departments of Rheumatology, Internal Medicine, Medical University of Graz, Graz
  - Rheumatology, Internal Medicine III, Medical University of Vienna, Vienna
  - Internal Medicine II, Hietzing Hospital, Vienna
- Germany (3):
  - Rheumatology, Charite, Berlin
  - Rheumatology, University of Düsseldorf, Düsseldorf
  - Internal Medicine III, University of Erlangen, Erlangen
- Netherlands (3):
  - Clinical Immunology, Groningen University Hospital, Groningen
  - Leiden University Medical Center, Netherlands, Leiden
  - Nephrology, University of Nymegen, Netherlands, Nijmegen

REFERENCES:
- [Background] Aringer M, Graninger WB, Steiner G, Smolen JS. Safety and efficacy of tumor necrosis factor alpha blockade in systemic lupus erythematosus: an open-label study. Arthritis Rheum. 2004 Oct;50(10):3161-9. doi: 10.1002/art.20576. PMID 15476222